CLINICAL TRIAL: NCT05402800
Title: Sexual Dysfunction in Infertile Women With PCOS Undergoing Fertility Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Bassiony Dabian, lecturer of obstetrics and gynecology, Cairo University
Other Study IDs: 12A34
Record Dates: First submitted 2022-05-29; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Sexual Dysfunction; PCOS
MeSH Terms: conditions — Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: FSFI questionnaire — The FSFI is a reliable test for the assessment of sexual function in women. The Arabic version of this test, was used. The FSFI is comprised of six domains (desire, arousal, lubrication, orgasm, satisfaction, and pain) with score ranges of 0 (or 1) to 5. The total FSFI score ranges from 2.0 to 36. The translated version of the FSFI test was used in this study. All questions in the FSFI questionnaire were explained by the physician one by one, and they were filled in a suitable and silent environment where patients could comfortably share such intimate information

SUMMARY:
Infertility, defined as the inability to become pregnant after one year of regular unprotected sexual intercourse. It is estimated that around 20 % of couples suffer from infertility with prevalence rates of infertility differing substantial among countries .

Sexual function in females is very complex and is affected by many factors. The prevalence of sexual dysfunction is higher in infertile patients compared to the normal population .

Whether sexual dysfunction is the cause or consequence of subfertility is difficult to establish. For instance, sexual dysfunction might result in decreased coital frequency compounding the issue of subfertility due to reduced exposure. On the other hand, the psychological pressure to get pregnant stemming from sex on demand could result in a reduction in enjoyment of sex aggravating sexual dysfunction. Indeed, situational sexual dysfunction and loss of a couple's intimacy may occur as a consequence of timed intercourse where focus for coitus is no longer pleasure but conception .

DETAILED DESCRIPTION:
Our work is an observational analytic cross-sectional study that included an Egyptian convenient sample of 186 females with primary infertility due to polycystic ovary syndrome.

Patients aged 18-35 were recruited from Kasr Al-Ainy Gynecology Clinic (Infertility Clinic) Medicine Hospital, Faculty of Medicine, Cairo University. They were diagnosed with primary infertility and polycystic ovary by Rotterdam criteria .

Patients with medical conditions (apart from PCOS complications like type II diabetes, obesity and metabolic syndrome) or receiving antidepressant therapy were excluded. Females with other causes of infertility associated with PCOS (e.g uterine factors, tubal factors) were not included. Patients with history of psychotic disorders or substance abuse were excluded. All patients approved to participate in the study and signed an informed consent to confirm this approval.

Intervention :

A- Gynecological Assessment :

Using Kasr Al Ainy infertility sheet that include clinical history taking of amenorrhea or oligomenorrhea. assessment of age years and type of infertility, medical history, surgical history, weight , height, history of hirsutism, ultrasound finding, speculum examination and hormonal profile including (FSH, LH, E2, Prolactin, TSH and progesterone) also history of any surgical intervention and type of fertility treatment were obtained . Vaginal ultrasound and speculum examination were done to every patient. PCOS was diagnosed using Rotterdam criteria based on identifying at least two of the following three features: oligo/anovulation , hyperandrogenism: clinical (hirsutism or male pattern alopecia) or biochemical (raised free androgen index or free testosterone) & polycystic ovaries on ultrasound (a follicle number per ovary of > 10).

Other etiologies must be excluded such as congenital adrenal hyperplasia, androgen secreting tumours, Cushing syndrome, thyroid dysfunction and hyperprolactinaemia .

Laboratory work up including :

1. LH/FSH ratio: Many women with PCOS have LH and FSH levels still within the 5-20 mlU/ml range, but their LH level is often two or three times that of the FSH level
2. Prolactin level: (1-20 ng/mL)
3. Estradiol level : (ranging from 20-400 pg/mL in healthy normal women)
4. TSH level : (normally 0.35- 5 μU/mL). TSH is checked to rule out other problems, such as an underactive or overactive thyroid, which often cause irregular or lack of periods and anovulation .

All blood samples (FSH-LH- E2 -PRL-TSH) were obtained at the second day of menstrual cycle in all women within the last six months before the interview

B-Data collection tool was a questionnaire completed through interviews in private meetings by the researcher. The questionnaire was composed of two parts: demographic characteristics and information about sexual relationship (such as frequency of sexual contacts per week, satisfaction with sexual and non-sexual relationships). Sexual dysfunction measurement were done by gynecologists/sexologists in infertility center on the basis of a diagnostic interview according to the Female Sexual Functioning Index (FSFI) The FSFI is a reliable test for the assessment of sexual function in women. The Arabic version of this test, was used. The FSFI is comprised of six domains (desire, arousal, lubrication, orgasm, satisfaction, and pain) with score ranges of 0 (or 1) to 5. The total FSFI score ranges from 2.0 to 36. The translated version of the FSFI test was used in this study. All questions in the FSFI questionnaire were explained by the physician one by one, and they were filled in a suitable and silent environment where patients could comfortably share such intimate information.

Analysis of data will be done by using SPSS ( statistical program for social science version 23 ) . Quantitative data will be statistically represented in terms of mean ± standard deviation (± SD) while categorical data will be represented as frequency and percentage. Comparison of quantitative data will be done using (Mann Whitney U ) test for independent samples while categorical data will be compared using ( Chi squared test ) or ( Fisher exact test ) when appropriate.

Correlation coefficient test will be used to rank different variables against each other where a probability value (p value) > 0.05 will be considered statistically insignificant , a probability value (p value) < 0.05 will be considered statistically significant & a probability value (p value) < 0.001 will be considered statistically highly significant.

ELIGIBILITY:
Inclusion Criteria:

1. Infertility .
2. PCOS.
3. Age from 18-35 years

Exclusion Criteria:

1. chronic medical condition previously associated with FSD (e.g. diabetes mellitus and cardiovascular diseases, such as hypertension) or using antidepressant medications.
2. Refusing participation in study.
3. Other causes of infertility

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients aged 18-35 were recruited from Kasr Al-Ainy Gynecology Clinic (Infertility Clinic) Medicine Hospital, Faculty of Medicine, Cairo University. They were diagnosed with primary infertility and polycystic ovary by Rotterdam criteria (8).
  Patients with medical conditions (apart from PCOS complications like type II diabetes, obesity and metabolic syndrome) or receiving antidepressant therapy were excluded. Females with other causes of infertility associated with PCOS (e.g uterine factors, tubal factors) were not included. Patients with history of psychotic disorders or substance abuse were excluded
Sampling Method: Non-Probability Sample
Enrollment: 186 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
prevalence of sexual dysfunction in PCOS | 6 months
  prevalence of sexual dysfunction in PCOS

SECONDARY OUTCOMES:
Risk factors for sexual dysfunction in PCO | 6 months
  Risk factors for sexual dysfunction in PCO
Relation of sexual dysfunction to different fertility treatments in PCO | 6 months
  Relation of sexual dysfunction to different fertility treatments in PCO

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy outpatient infertility clinic, Cairo, Egypt

REFERENCES:
- [Background] World Health Organization. Report of a WHO meeting. In: Vayena E, Rowe PJ, Griffin PD, editors. Current practices and controversies in assisted reproduction. Geneva: Byword Editorial Consultants; 2002. p. 1-396
- [Background] Fassino S, Piero A, Boggio S, Piccioni V, Garzaro L. Anxiety, depression and anger suppression in infertile couples: a controlled study. Hum Reprod. 2002 Nov;17(11):2986-94. doi: 10.1093/humrep/17.11.2986. PMID 12407062
- [Background] Malin M, Hemmink E, Raikkonen O, Sihvo S, Perala ML. What do women want? Women's experiences of infertility treatment. Soc Sci Med. 2001 Jul;53(1):123-33. doi: 10.1016/s0277-9536(00)00317-8. PMID 11380158
- [Background] Ercan CM, Coksuer H, Aydogan U, Alanbay I, Keskin U, Karasahin KE, Baser I. Sexual dysfunction assessment and hormonal correlations in patients with polycystic ovary syndrome. Int J Impot Res. 2013 Jul-Aug;25(4):127-32. doi: 10.1038/ijir.2013.2. Epub 2013 Feb 14. PMID 23407282
- [Background] Keye WR Jr. Psychosexual responses to infertility. Clin Obstet Gynecol. 1984 Sep;27(3):760-6. doi: 10.1097/00003081-198409000-00024. PMID 6488617
- [Background] Rotterdam ESHRE/ASRM-Sponsored PCOS Consensus Workshop Group. Revised 2003 consensus on diagnostic criteria and long-term health risks related to polycystic ovary syndrome. Fertil Steril. 2004 Jan;81(1):19-25. doi: 10.1016/j.fertnstert.2003.10.004. PMID 14711538